CLINICAL TRIAL: NCT05867511
Title: A Pilot Feasibility Study to Promote Physical Activity Motivation in Cardiovascular Disease Patients
Brief Title: A Study to Promote Physical Activity Motivation in Cardiovascular Disease Patients
Acronym: iPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudio Nigg (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Claudio Nigg, Prof. Dr. Claudio Nigg, University of Bern
Organization: University of Bern (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-02500
Record Dates: First submitted 2023-03-07; First posted 2023-05-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Health behavior change; Physical activity; Sedentary behavior; App based intervention; Transtheoretical model; Habit formation
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The study is a one-armed pilot 8-week tailored intervention with a pre-post-design, as well as an intensive-longitudinal design with weekly measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): This Group will be using the iPAL App for 8 Weeks
  Interventions: Behavioral: iPAL App

INTERVENTIONS:
Behavioral: iPAL App — The intervention will have a duration of eight weeks. It is theory-based, will be delivered to participants' smartphones via the study app (except components 5 and 6), and comprises the following components:
  1. Theory-based individualized feedback.
  2. Self-generated motivational messages.
  3. Motivation for habit formation through push messages.
  4. Motivational images and videos that participants handed in or selected will be sent to them through the app.
  5. Study-specific social media groups. Participants will be offered the option to participate in study-specific social media groups.
  6. Posting motivational stories. A story of a person, who successfully changed his or her lifestyle to be more physically active and/or less sedentary, will be posted once a week in the study-specific social media groups.

SUMMARY:
This study investigates the feasibility of an app based intervention, which uses questionnaires and personalized motivational messages to achieve change in physical activity and sedentary behaviour of cardiovascular patients. The questionnaires and messages are based on behaviour change theories, such as the transtheoretical model. The intervention will take place over eight weeks. One week before and during the last week, physical activity will be measured via accelerometers. A comprehensive questionnaire will be given before and at the end of the intervention and Feasibility measures will be evaluated at the end as well, including an optional qualitative interview with the participants.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death and disability worldwide. They are mainly caused by lifestyle risk factors, such as physical inactivity, which is also the fourth leading risk factor for mortality. Regular physical activity is crucial for the prevention and treatment of cardiovascular diseases. Nevertheless, success in achieving long-term adherence to physical activity recommendations after an acute cardiac event or even after exercise-based cardiac rehabilitation is rather low. Furthermore, even though most research has focused on physical activity, engaging in reduced amounts of sedentary behavior is also crucial, as it represents an important cardiovascular risk even after adjusting for physical activity. Health behavior change theories, such as the transtheoretical model, and empirical evidence highlight the importance of motivation and motivational factors in the behavior maintenance or change process. Thus, the main goal of the present study is to assess preliminary effectiveness of an intervention mostly based on the transtheoretical model to promote cardiovascular patients' motivation to be physically active and to engage in reduced amounts of sedentary behavior. Most intervention components will be delivered digitally to the participants' smartphones via a study specific app. Furthermore, weekly questionnaires allow the investigators' to individualize the intervention components and investigate associations not only between-subjects, but also within-subjects over time, which is essential and has been neglected in the literature. The primary objective is to assess study feasibility.

ELIGIBILITY:
Inclusion criteria:

* Cardiovascular disease patients
* Participating in cardiovascular rehabilitation OR having received the recommendation from a cardiologist to participate in cardiovascular rehabilitation and having refused
* Signing the informed consent form
* Owning a smartphone with internet access

Exclusion criteria:

* Age under 18 years
* Having a contraindication for physical activity
* Existing or suspected non-fulfilment of the participation requirements
* Inability to follow the procedures of the study (e.g., by not speaking German, being unable to read or write, or severe cognitive impairment)
* Being in palliative care
* Being pregnant
* Having an assisted living situation
* Stroke patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of approached patients included | Approx. 5 Months
  The goal is to include at least 10% of approached patients.
Dropout rate | Participants can dropout at any time during the study (during 9 weeks for each participant)
  The goal is that the dropout rate is lower than 50%
Completion of study assessments | Participants may fill out study questionnaires weekly during the 8-week intervention or not.
  The goal is that, on average participants complete at least 4 out of 9 of the questionnaires of the study. Excluding dropouts.

SECONDARY OUTCOMES:
Overall satisfaction | Last questionnaire of the study for each participant (post questionnaire right after the 8 intervention weeks; 9 weeks after study start)
  Overall satisfaction with the intervention will be assessed via the post-questionnaire based on the Questionnaire to Measure Patient Satisfaction (in German: "Fragebogen zur Messung der Patientenzufriedenheit"; ZUF-8; Attkisson & Zwick, 1982) as part of study feasibility. Each of the nine item based on the ZUF-8 is rated on a 0 to 3 Likert-scale (or 3 to 0 for reversed items) with higher rating indicating higher satisfaction. Items are summed up to build a score, which ranges from 0 to 27.
Usability | Last questionnaire of the study for each participant (post questionnaire right after the 8 intervention weeks; 9 weeks after study start)
  Usability will be assessed via the post-questionnaire based on System Usability Scale (Brooke, 1996) as part of study feasibility. The ten items are rated on a six point Likert-scale coded from 0 to 5 with some items having to be reversed. A score is built as the sum of the items (after reversing the pertinent ones). Thus, scores range from 0 to 50 with higher scores indicating better usability.
Engagement | Last questionnaire of the study for each participant (post questionnaire right after the 8 intervention weeks; 9 weeks after study start)
  Engagement will be assessed via the post-questionnaire based on Digital Behaviour Change Interventions Engagement Scale (Perski et al., 2020) as part of study feasibility. The eight items are rated on a seven point Likert-scale from "not at all" (1) to "extremely" (7). After reversing the pertinent items, an overall engagement score can be built as the mean of the items. Thus, scores range from 1 to 7 with higher scores indicating greater engagement.
Satisfaction with the specific intervention components | Last questionnaire of the study for each participant (post questionnaire right after the 8 intervention weeks; 9 weeks after study start)
  Satisfaction for each intervention component will be assessed via the post-questionnaire based on two items from the Questionnaire to Measure Patient Satisfaction (ZUF-8; Attkisson & Zwick, 1982) for each intervention component as part of study feasibility. Items are rated on a Likert-scale coded from 0 to 3. Scores are built as the sum of the two items. Thus, satisfaction scores range from 0 to 6 for each intervention component with higher scores indicating higher satisfaction.
Needs assessment | Last questionnaire of the study for each participant (post questionnaire right after the 8 intervention weeks; 9 weeks after study start)
  Needs assessment for personal contact will be assessed via the post-questionnaire roughly based on the satisfaction, usability and engagement scales mentioned above and as part of study feasibility. Items are rated on a 5-point Likert scale from "not agreeing at all" (1) to "agreeing completely" (5). After reversing the pertinent items, an overall score can be built as the mean of the items. Thus, scores range from 1 to 5 with higher scores indicating a higher need for personal contact.
Motivation | Weekly right before, during and right after the 8-week intervention for each participant.
  Motivation for physical activity will be measured by Situational Motivation Scale (SIMS) at the pre- and post-questionnaires as well as in the shortened form during the weekly questionnaires (4 items; short form not validated). The SIMS includes 16 items rated on a 7-point Likert-scale ranging from "not at all in agreement " (1) to "completely in agreement" (7). Four items form each of the following subscales: intrinsic motivation, identified regulation, external regulation, and amotivation. A score for each subscale is built as the mean of the four items (or, in the case of the weekly questionnaire, the rating of the single item directly). Thus, scores range from 1 to 7 with higher scores indicating a higher motivation.
Stage of change | Weekly right before, during and right after the 8-week intervention for each participant.
  Further indicators of motivation will be the motivational factors of the transtheoretical model (TTM) based on validated items from Lee et al. (2001) and Paxton et al. (2008). Stage of change will be assessed using one question with five answer alternatives at every questionnaire. The answer directly indicates the stage the person is at (precontemplation, contemplation, preparation, action, or maintenance). The question will be included once for physical activity motivation and once for sedentary behavior motivation (the latter also based on Han et al., 2017).
Processes of change | Weekly right before, during and right after the 8-week intervention for each participant.
  The 5-factor model of processes of change from the transtheoretical model for physical activity will be assessed with 22 items in the pre- and post-, and 5 items in the weekly questionnaires based on Paxton et al. (2008). All items are rated on a 5-point Likert-scale from 1 to 5 and a score for each of the five factors is built as the average of the corresponding items. Thus, scores range from 1 to 5. Higher scores indicate a more frequent use of each process of change.
Decisional balance | Weekly right before, during and right after the 8-week intervention for each participant.
  Decisional balance (as a factor of the transtheoretical model for physical activity) will be assessed with 13 items in the pre- and post-, and 4 items in the weekly questionnaires (based on Paxton et al., 2008). Items are rated on a 5-point Likert-scale from 1 to 5. Two scores are built, one for pros and one for cons, as the mean of the corresponding items. Thus, scores range from 1 to 5 with higher scores indicating more importance of the pros or cons. Decisional balance for sedentary behavior will be measured as well with 16 items in the pre- and post-, and with four items in the weekly questionnaires (based on Han et al., 2017; Paxton et al., 2008). Scoring is exactly the same as for decisional balance for physical activity.
Self-efficacy | Weekly right before, during and right after the 8-week intervention for each participant.
  Self-efficacy (as a variable of the transtheoretical model) will be measured once for physical activity and once for sedentary behavior using 7 items in the pre- and post-, and 1 item in the weekly questionnaires (based on Paxton et al., 2008; Han et al., 2017). Items are rated on a 5-poin Likert-scale ranging from 1 to 5. A score is built by averaging the items. Thus, scores range from 1 to 5 with higher scores indicating higher self-efficacy.
Temptation | Weekly right before, during and right after the 8-week intervention for each participant.
  Temptation (as a factor of the transtheoretical model for physical activity) will be assessed with seven items during the pre- and post-questionnaires and- with two items during the weekly questionnaires (based on Paxton et al.; 2008). The items are rated on a continuous scale from 0% to 100%. A score for affect and one for competing demands is built as the average of the corresponding items. Thus, scores range from 0% to 100% with higher scores indicating higher temptation.
Social support | Weekly right before, during and right after the 8-week intervention for each participant.
  self reported social support pertaining physical activity will be measured based on items by Rackow et al., 2017 (not validated, but based on previous literature). Single items are used in each questionnaire to measure the following subscales: quantity of practical social support, quality of practical social support, quantity of emotional social support, and quality of emotional social support. Items are rated on 6-point Likert scales ranging from 0 to 5. The single ratings for quality already represent a score for quantity of practical and emotional support, accordingly. Thus, scores range from 0 to 5 with higher scores indicating a higher quantity of social support. In order to take quality into account, scores ca be built by multiplying the quantity with the quality item once for practical support and ince for social support. These scores would range from 0 to 25 with higher scores indicating more and better support.
Habit | Weekly right before, during and right after the 8-week intervention for each participant.
  habit will be measured via self-report based on validated Self-Report Habit Index (Gardner et al., 2012). The four items are rated on a 5-point Likert-scale from 0 to 4. A score is built by averaging the items. Thus, scores range from 0 to 4 with higher values representing a higher automaticity (a stronger habit). The scale will be applied once for physical activity, once for sedentary behavior, and once for a reduction of sedentary behavior.
Affect | Weekly right before, during and right after the 8-week intervention for each participant.
  positive and negative affect will be assessed with a validated scale by Krohne et al.(1996), the short and German version of the Positive and Negative Affect Schedule. Ten items are rated on a 5-point Likert-scale from 0 to 4, five items measure positive and five negative affect. Scores are built as the mean of the corresponding items for positive and negative affect. Thus, scores range from 0 to 4 with higher values indicating higher levels of positive/negative affect.
Self reported health-related quality of life | Weekly right before, during and right after the 8-week intervention for each participant.
  Self reported health-related quality of life assessed with the validated instrument MacNew Heart Disease Health-Related Quality of Life Questionnaire (MacNew; Höfer et al., 2004). Originally, the scale includes 27 items rated on a 7-point Likert-scale from 1 to 7. However, we excluded one item as recommended in the literature due to very low response rate in previous research. A global quality of life score can be built by averaging the remaining 26 items. Furthermore, scores for a physical, an emotional and a social subscale can be built by averaging the corresponding items. (We recommend following the factorial structure proposed by Bermudez et al. (2022) given that the original structure has shown some issues.) Thus. all scores range from 1 to 7 with higher scores indicating higher quality of life.
Physical activity | Self-report: Weekly right before, during and right after the 8-week intervention. Device-based: during the 8 days before and the last 7 days of the intervention.
  Self reported physical activity will be assessed with an adapted version of the Godin-Shepherd Leisure-Time Physical Activity Questionnaire (Godin, 2011). Participants indicate on how many of the last seven days and for how many minutes per day they engaged in each type of physical activity (light, moderate, vigorous). Scores for each type of activity are built by multiplying the amount of days with the amount of minutes. Another score will be built for moderate-to-vigorous physical activity in minutes per week by adding the score of vigorous und moderate activity. Thus, higher activity scores indicate more minutes per week engaged in each type of activity. Device based assessment of physical activity will be done with a triaxial accelerometer. As with the self-report outcomes will me light, moderate, vigorous and moderate-to-vigorous physical activity per week in minutes (with higher scores indicating more minutes engaged in each activity per week).
Sedentary behaviour | Self-report: Weekly right before, during and right after the 8-week intervention. Device-based: during the 8 days before and the last 7 days of the intervention.
  Self reported physical activity will be assessed with the Measure of Older Adults' Sedentary Time (MOST; Gardiner et al. 2011). Participants indicate on how many of the last seven days and for how many minutes per day they engaged in seven different sedentary activities. A score is built by multiplying the amount of days with the amount of minutes for each sedentary activity and summing them up. Thus, scores represent amount of sedentary time per week in minutes (with higher scores indicating more sedentary time). Device based assessment of sedentary behavior will be done with a triaxial accelerometer. Outcome will be sedentary time in minutes per week (thus, higher scores indicate more sedentary time).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Nigg, PhD, Principal Investigator — University of Bern
Locations (1):
- Institute of Sport Science, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Bolger, N., & Laurenceau, J. P. (2013). Intensive longitudinal methods: An introduction to diary and experience sampling research. Guilford Press.
- [Background] Brooke, J. (1996). SUS-A quick and dirty usabiliy scale. Usability Evaluation in Industry, 189(194), 4-7.
- [Background] Dolansky MA, Stepanczuk B, Charvat JM, Moore SM. Women's and men's exercise adherence after a cardiac event. Res Gerontol Nurs. 2010 Jan;3(1):30-8. doi: 10.3928/19404921-20090706-03. Epub 2010 Jan 27. PMID 20128541
- [Background] Gardner B, Abraham C, Lally P, de Bruijn GJ. Towards parsimony in habit measurement: testing the convergent and predictive validity of an automaticity subscale of the Self-Report Habit Index. Int J Behav Nutr Phys Act. 2012 Aug 30;9:102. doi: 10.1186/1479-5868-9-102. PMID 22935297
- [Background] Greaney ML, Riebe D, Ewing Garber C, Rossi JS, Lees FD, Burbank PA, Nigg CR, Ferrone CL, Clark PG. Long-term effects of a stage-based intervention for changing exercise intentions and behavior in older adults. Gerontologist. 2008 Jun;48(3):358-67. doi: 10.1093/geront/48.3.358. PMID 18591361
- [Background] Halloway S, Wilbur J, Schoeny ME, Semanik PA, Marquez DX. Combined Effects of Sedentary Behavior and Moderate-to-Vigorous Physical Activity on Cardiovascular Health in Older, Community-Dwelling Latinos. J Aging Phys Act. 2016 Apr;24(2):296-304. doi: 10.1123/japa.2015-0096. Epub 2015 Oct 6. PMID 26439328
- [Background] Höfer, S., Benzer, W., Brandt, D., Laimer, H., Schmid, P., Bernardo, A [Arthur], & Oldridge, N. B. (2004). MacNew Heart Disease Lebensqualitätsfragebogen nach Herzinfarkt. Zeitschrift Für Klinische Psychologie Und Psychotherapie, 33(4), 270-280. https://doi.org/10.1026/1616-3443.33.4.270
- [Background] Khan MA, Hashim MJ, Mustafa H, Baniyas MY, Al Suwaidi SKBM, AlKatheeri R, Alblooshi FMK, Almatrooshi MEAH, Alzaabi MEH, Al Darmaki RS, Lootah SNAH. Global Epidemiology of Ischemic Heart Disease: Results from the Global Burden of Disease Study. Cureus. 2020 Jul 23;12(7):e9349. doi: 10.7759/cureus.9349. PMID 32742886
- [Background] Krohne, H. W., Egloff, B., Kohlmann, C.-W., & Tausch, A. (1996). Untersuchungen mit einer deutschen Version der Positive and Negative Affect Schedule (PANAS). Diagnostica, 42(2), 139-156.
- [Background] Lee RE, Nigg CR, DiClemente CC, Courneya KS. Validating motivational readiness for exercise behavior with adolescents. Res Q Exerc Sport. 2001 Dec;72(4):401-10. doi: 10.1080/02701367.2001.10608976. PMID 11770789
- [Background] Nigg, C. R [C. R.], & Riebe, D. (2002). The Transtheoretical Model: Research review of exercise behavior and older adults. In P. Burbank & D. Riebe (Eds.), Promoting exercise and behavior change in older adults: interventions with the Transtheoretical Model (pp. 147- 180). Springer Publishing Company.
- [Background] Paxton RJ, Nigg CR, Motl RW, McGee K, McCurdy D, Matthai CH, Dishman RK. Are constructs of the transtheoretical model for physical activity measured equivalently between sexes, age groups, and ethnicities? Ann Behav Med. 2008 Jun;35(3):308-18. doi: 10.1007/s12160-008-9035-x. Epub 2008 Jul 8. PMID 18607667
- [Background] Perski O, Blandford A, Garnett C, Crane D, West R, Michie S. A self-report measure of engagement with digital behavior change interventions (DBCIs): development and psychometric evaluation of the "DBCI Engagement Scale". Transl Behav Med. 2020 Feb 3;10(1):267-277. doi: 10.1093/tbm/ibz039. PMID 30927357
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Rackow, P., Berli, C., Lüscher, J., Luszczynska, A., & Scholz, U. (2017). Emotional or instrumental support? Distinct effects on vigorous exercise and affect. Psychology of Sport and Exercise, 33, 66-74. https://doi.org/10.1016/j.psychsport.2017.07.011
- [Background] ter Hoeve N, Huisstede BM, Stam HJ, van Domburg RT, Sunamura M, van den Berg-Emons RJ. Does cardiac rehabilitation after an acute cardiac syndrome lead to changes in physical activity habits? Systematic review. Phys Ther. 2015 Feb;95(2):167-79. doi: 10.2522/ptj.20130509. Epub 2014 Oct 2. PMID 25278337
- [Background] WHO. (2017, August). Global strategy on diet, physical activity and health: Physical activity. http://www.who.int/dietphysicalactivity/pa/en/
- [Background] WHO. (2020, December 9). The top 10 causes of death. https://www.who.int/news-room/factsheets/detail/the-top-10-causes-of-deat
- [Background] Godin, G. (2011). The Godin-Shephard leisure-time physical activity questionnaire. The Health & Fitness Journal of Canada, 4(1), 18-22.
- [Background] Gardiner PA, Clark BK, Healy GN, Eakin EG, Winkler EA, Owen N. Measuring older adults' sedentary time: reliability, validity, and responsiveness. Med Sci Sports Exerc. 2011 Nov;43(11):2127-33. doi: 10.1249/MSS.0b013e31821b94f7. PMID 21448077
- [Background] Han H, Pettee Gabriel K, Kohl HW 3rd. Application of the transtheoretical model to sedentary behaviors and its association with physical activity status. PLoS One. 2017 Apr 27;12(4):e0176330. doi: 10.1371/journal.pone.0176330. eCollection 2017. PMID 28448531
- [Background] Bermudez T, Bierbauer W, Scholz U, Hermann M. Depression and anxiety in cardiac rehabilitation: differential associations with changes in exercise capacity and quality of life. Anxiety Stress Coping. 2022 Mar;35(2):204-218. doi: 10.1080/10615806.2021.1952191. Epub 2021 Jul 16. PMID 34269151